CLINICAL TRIAL: NCT02540408
Title: COPD in Dairy Farmers: Screening, Characterization and Constitution of a Cohort. The BALISTIC Study
Brief Title: Detection and Characterization of COPD in Dairy Farmers
Acronym: BALISTIC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P-2011-119
Record Dates: First submitted 2013-08-29; First posted 2015-09-04 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Environmental Exposure
Keywords: Occupational COPD; Pathophysiology; Exercise limitation; Pulmonary hyperinflation; Arterial stiffness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum for further analyses
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- presence of COPD: COPD patients are defined according to the results of a spirometry

SUMMARY:
A pilot study from the investigators group suggests that the prevalence of chronic obstructive pulmonary disease (COPD) among dairy farmers is higher than in the general population. Most characteristics of COPD in dairy farmers (smoking habits, dyspnoea, quality of life, lung function, bronchial exhaled nitric oxide, systemic inflammation, arterial stiffness and exercise capacity) are largely unknown. Although immunization against organic dusts is suspected, the pathophysiology of COPD in dairy farmers is also unknown.

This study therefore aims at (i) comparing the prevalence of COPD in dairy farmers and in subjects without any occupational exposure (control arm) through a vast COPD detection program in the Franche-Comté region; (ii) comparing several characteristics (smoking habits, dyspnoea, quality of life, lung function, bronchial exhaled nitric oxide, systemic inflammation, arterial stiffness and exercise capacity) between dairy farmers with COPD and patients with COPD without any occupational exposure; (iv) identifying etiological factors of COPD in dairy farmers (comparison of exposure and specific immunoglobulin E between dairy farmers with COPD and dairy farmers with normal pulmonary function tests); and (v) constituting a cohort of COPD patients and control subjects for further longitudinal studies.

Data from selected patients (either current or former smokers) with mild COPD and from matched controls will also be analyzed in an ancillary study which objectives are to compare exercise tolerance, ventilatory constraints on tidal volume expansion and dyspnoea between asymptomatic mild COPD subjects, symptomatic mild COPD and healthy controls.

DETAILED DESCRIPTION:
2000 dairy workers and 2000 subjects without any occupational exposure, all aged 40 to 74 years, will take part to a COPD screening program (spirometry and bronchodilation test) between September 2011 and October 2014.

Subjects with COPD and healthy matched controls will attend a second visit. If needed, COPD subjects will be asked to stop any respiratory related medication such as short and long acting bronchodilators 72 hours prior to the visit. All subjects will complete several questionnaires (quality of life, respiratory symptoms, smoking habits,…). A complete medical history will be collected, and a blood sample will be taken. Subjects thereafter will complete arterial stiffness measurement, exhaled nitric oxide and pulmonary function testing pre- and 30-min post-bronchodilator. A symptom-limited incremental cycle exercise test will be performed on the same day, at least 6 hours after the bronchodilator test and at least 4 hours after the meal.

Exposure to organic dusts will be quantified through analyze of electrostatic wipes left at subjects' homes for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* subject aged 40-74 years
* either dairy farmer or unexposed to any occupational risk factor for COPD

Exclusion Criteria:

* COPD in GOLD stage 4
* pregnancy
* treatment with systemic corticosteroids
* established diagnosis of asthma
* established diagnosis of bronchiectasis
* established diagnosis of allergic alveolitis

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD patients will be defined according to the GOLD criteria (post-bronchodilator FEV1/FVC ratio<70%).
  Healthy subjects must have pre-bronchodilator FEV1/FVC ratio >75% and pre-bronchodilator FEV1 >95% of predicted value.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
prevalence of COPD in dairy farmers and in unexposed subjects | 3-year

SECONDARY OUTCOMES:
comparison of smoking habits between dairy farmers with COPD and unexposed COPD | 4-year
comparison of dyspnoea between dairy farmers with COPD and unexposed COPD | 4-year
  , quality of life, lung function, bronchial exhaled nitric oxide, systemic inflammation, arterial stiffness and exercise capacity
comparison of lung function between dairy farmers with COPD and unexposed COPD | 4-year
comparison of bronchial exhaled nitric oxide between dairy farmers with COPD and unexposed COPD | 4-year
comparison of systemic inflammation between dairy farmers with COPD and unexposed COPD | 4-year
comparison of arterial stiffness between dairy farmers with COPD and unexposed COPD | 4-year
comparison of exercise capacity between dairy farmers with COPD and unexposed COPD | 4-year
comparison of exposure to organic dusts between dairy farmers with and without COPD | 3-year
comparison of immunization to organic dusts between dairy farmers with and without COPD | 3-year

OTHER OUTCOMES:
comparison of dyspnoea between asymptomatic mild COPD subjects, symptomatic mild COPD and healthy controls | 2-year
  the magnitude of their perceived breathing discomfort at rest, at the middle of warm up, every 2-minute during exercise, and at peak exercise is rated by pointing to the 10-point Borg scale
comparison of exercise tolerance dyspnoea between asymptomatic mild COPD subjects, symptomatic mild COPD and healthy controls | 2-year
comparison of ventilatory constraints on tidal volume expansion between asymptomatic mild COPD subjects, symptomatic mild COPD and healthy controls | 2-year
  In the relationship between tidal volume (VT) and ventilation (V'E), there is an inflection point beyond which almost no further change in VT is possible despite a continued increase in V'E. This inflection in the VT response marks the point were dyspnoea sharply raises because of mechanical constraints on VT expansion. This inflection point is determined for each patient by analyzing individual Hey plot.
cardiovascular risk in COPD patients either never-smokers or current/former smokers | 3-year
  comparison of pulse wave velocity between smoking and non-smoking COPD

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Degano, MD, PhD, Principal Investigator — CHU Besançon; Jean-Charles Dalphin, MD, PhD, Study Chair — CHU Besançon
Locations (1):
- CHU Jean Minjoz, Besançon, France

REFERENCES:
- [Background] Degano B, Bouhaddi M, Laplante JJ, Botebol M, Annesi-Maesano I, Marescaux A, Roux P, Thaon I, Wolf JP, Regnard J, Dalphin JC. [COPD in dairy farmers: screening, characterization and constitution of a cohort. The BALISTIC study]. Rev Mal Respir. 2012 Nov;29(9):1149-56. doi: 10.1016/j.rmr.2012.08.007. Epub 2012 Oct 15. French. PMID 23200591
- [Derived] Veil-Picard M, Soumagne T, Vongthilath R, Annesi-Maesano I, Guillien A, Laurent L, Andujar P, Roche N, Jouneau S, Cypriani B, Laplante JJ, Degano B, Dalphin JC. Is atopy a risk indicator of chronic obstructive pulmonary disease in dairy farmers? Respir Res. 2019 Jun 17;20(1):124. doi: 10.1186/s12931-019-1082-2. PMID 31208466